CLINICAL TRIAL: NCT03276741
Title: Unrestricted Low Fat, Low Residue Oral Intake During Labor: A Randomized Controlled Study
Brief Title: Oral Intake During Labor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit to enrollment target
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeanette Anderson, Branch Chief, Provision of Inpatient Nursing Care, David Grant U.S. Air Force Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FDG20170006H
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Labor Complication; Food Aspiration; Complication of Anesthesia; Satisfaction
Keywords: labor; anesthesia; oral intake; maternal satisfaction; newborn complications
MeSH Terms: conditions — Obstetric Labor Complications; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: quantitative, randomized experimental design study
Who Masked: Outcomes Assessor
Masking Description: Personal identification removed (use of personal identification code)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine care during labor (authorized clear liquid diet).
- Experimental Group (Active Comparator): Patients in the experimental group will have a gastric soft/bland diet available, which will include lean protein, fruits, vegetables, and low-fat dairy. This will be ordered in the electronic medical record (EMR) and is a standard "non-select meal," referred to as a gastric/soft bland diet that is not based on patient's preferred menu selections.
  Interventions: Dietary Supplement: gastric soft/bland diet

INTERVENTIONS:
Dietary Supplement: gastric soft/bland diet — Patients in the experimental group will have a gastric soft/bland diet available.
  Arms: Experimental Group

SUMMARY:
A randomized clinical trial (RCT) to evaluate the impact of unrestricted low fat, low residue oral intake during labor on maternal and neonatal outcomes as well as maternal satisfaction.

DETAILED DESCRIPTION:
This study is a quantitative, randomized experimental design study to determine the impact of unrestricted low fat, low residue oral intake during labor on the indicated outcome variables and patient satisfaction. The comparison group will continue standard care of being allowed a clear liquid during active labor (≥6cm dilation), while the experimental group would be allowed to self-regulate oral intake with a low fat, low residue diet during active labor.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty and Department of Defense (DoD) beneficiary Pregnant women 18 years of age and older
* 37 weeks gestation or greater at time of admission
* singleton fetus
* cephalic presentation
* who plan to labor/deliver at DGMC (military beneficiaries).

Exclusion Criteria:

* Morbid/severe obesity (pre-pregnancy BMI ≥40 kg/m2
* diabetes
* hypertension (to include pre-eclampsia or eclampsia)
* previous cesarean section
* uncontrolled gastroesophageal reflux disease (GERD) (symptomatic with medication)
* past history or current diagnosis of hyperemesis gravidarum
* food allergies to any items contained in the gastric/soft bland diet
* patients utilizing nitrous oxide for labor analgesia (should this treatment be available at DGMC)
* Difficult airway as defined by the anesthesia staff.
* Mallampati score 3 or 4
* Thyroid mental distance less than 7 cm or 3 finger breaths
* Mouth opening less than 3 finger breaths
* Short thick neck, Micrognathia
* Further indications as determined by the anesthesia provider doing the anesthesia preoperative assessment (pregnancy in and of itself will not be considered a disqualification due to airway changes during labor)" in order to define difficult airway per anesthesia.
* Under age 18
* Additional clinical risk factors as determined by the care provider

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study includes pregnant women
Enrollment: 126 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-01-11 (Actual)

PRIMARY OUTCOMES:
Nausea | active labor (6cm or greater dilation) through delivery of the infant
  # episodes
Vomiting | active labor (6cm or greater dilation) through delivery of the infant
  # episodes
Duration of labor | active labor (6cm or greater dilation) through delivery of the infant
  #hours/minutes
Mode of delivery | at birth
  cesarean section, operative vaginal delivery, spontaneous vaginal delivery
Aspiration | active labor (6cm or greater dilation) through delivery of the infant
  # episodes
Newborn APGAR Score | 5 min of life
  < 7
Maternal Satisfaction | active labor (6cm or greater dilation) through delivery of the infant
  open ended survey question

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette M Anderson, MSN, Principal Investigator — David Grant Medical Center
Locations (1):
- USAF David Grant Medical Center, Travis Air Force Base, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03276741/ICF_000.pdf